CLINICAL TRIAL: NCT00139971
Title: Phase III Study of Gemcitabine Compared With UFT in Patients With Completely Resected Pathological Stage IB-IIIa Non Small Cell Lung Cancer
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: West Japan Thoracic Oncology Group (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: WJTOG0101
Record Dates: First submitted 2005-08-30; First posted 2005-08-31 (Estimated); Last update posted 2006-01-06 (Estimated); Status verified 2005-08

CONDITIONS: Lung Cancer
MeSH Terms: conditions — Lung Neoplasms | interventions — Gemcitabine; Tegafur

INTERVENTIONS:
Drug: gemicitabine 1000mg/m2, day1 and day 8, every 3 week, 6
Drug: UFT 250mg/m2, daily for 1 year

SUMMARY:
To estimate the efficacy of Gemcitabine monotherapy compared to UFT as the post operative adjuvant chemotherapy for completely resected non-small cell lung cancer.

ELIGIBILITY:
Inclusion Criteria:

1. completely resected non small cell lung cancer
2. no prior anti cancer treatment for thoracic malignancy exept for this operation
3. pathological stage IB, II, and stage IIIA with only one station of n2 disease
4. PS 0-1
5. age 20-75
6. adequate organ function for chemotherapy
7. written informed consent

Exclusion Criteria:

1. small cell lung cancer or low grade malignancy of lung cancer
2. incomplete resection
3. apparent interstitial pneumonitis at chest rentogenogram
4. inadequate condition for chemotherapy

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 600
Dates: Start 2001-12

PRIMARY OUTCOMES:
5 year survival rate

SECONDARY OUTCOMES:
Disease free survival

CONTACTS AND LOCATIONS:
Overall Officials: Hirohito Tada, MD, Principal Investigator — West Japan Thoracic Oncology Group
Locations (1):
- Osaka City General Hospital, Osaka, Osaka, Japan

REFERENCES:
- See also: Related Info — http://www.wjtog.org/